CLINICAL TRIAL: NCT03516123
Title: A Phase I, Open Label, Multiple Dose, Dose Escalation and Expansion Study to Investigate the Safety, Tolerability, PK and Antitumor Activities of the MEK Inhibitor CS3006 in Subjects with Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of CS3006 in Subjects with Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS3006-101
Record Dates: First submitted 2018-04-22; First posted 2018-05-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2020-03

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — MEK inhibitor I

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CS3006 (Experimental): Participants will receive CS3006 orally at specified dose on specified days
  Interventions: Drug: CS3006

INTERVENTIONS:
Drug: CS3006 — In the dose escalation part, the dose levels will be escalated following a modified 3+3 dose escalation scheme.
  In the dose expansion part, participants will receive CS3006 at specified dose level(s).
  Other Names: MEK inhibitor

SUMMARY:
This is a multicenter, open label, dose escalation & expansion phase I study to evaluate the clinical safety, tolerability, PK, and preliminary efficacy of CS3006.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histologically or cytologically confirmed advanced or metastatic solid tumor(s) for which no effective standard therapy is available or tolerable.
2. ECOG performance status of 0 or 1.
3. Life expectancy ≥12 weeks.
4. Able to swallow and retain oral medication.
5. Subjects must have adequate organ function.
6. Use of effective contraception.

Exclusion Criteria:

1. Subjects receiving anti-cancer therapy at the time of enrollment.
2. Subjects who had prior chemotherapy, targeted therapy, immunotherapy or any other systemic anti-cancer treatment, within 14 days prior to the first dose of CS3006 or who has not recovered from adverse events due to a prior therapy.
3. Receipt of any prior therapy with a MEK inhibitor.
4. Use of any investigational anti-cancer drug within 28 days before the first dose of CS3006.
5. Current use of a prohibited medication or use during treatment of CS3006.
6. Current use of warfarin.
7. Any condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of drugs.
8. History of retinal vein occlusion (RVO) or central serous retinopathy (CSR).
9. Visible retinal pathology as assessed by ophthalmologic exam.
10. Intraocular pressure > 21mm Hg as measured by tomography.
11. Glaucoma diagnosed within one month prior to the first dose of CS3006.
12. Known brain metastasis or other CNS metastasis that is either symptomatic or untreated.
13. Primary malignancy of CNS.
14. Evidence of severe or uncontrolled systemic diseases.
15. Subjects with clinically significant cardiovascular disease.
16. QTc interval >= 450 msecs for male or >= 470 msecs for female
17. Known history of HIV.
18. Subjects with active Hepatitis B or C infection
19. History of immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to CS3006.

For more information regarding trial participation, please contact at cstonera@cstonepharma.com

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | From the day of first dose to 30 days after last dose of CS3006

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Huang, Study Director — CStone Pharmaceuticals
Locations (1):
- St Vincent's hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No